CLINICAL TRIAL: NCT02081456
Title: The Effects of Soft Tissue Mobilization Versus Therapeutic Ultrasound for Subjects With Neck and Arm Pain With Evidence of Neural Mechanical Sensitivity: A Randomized Clinical Trial
Brief Title: Soft Tissue Mobilization Versus Therapeutic Ultrasound for Subjects With Neck and Arm Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emilio J Puentedura, PT, DPT, PhD (Other)
Responsible Party: Sponsor-Investigator, Emilio J Puentedura, PT, DPT, PhD, Co-Principal Investigator, University of Nevada, Las Vegas
Organization: University of Nevada, Las Vegas (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-242
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic Ultrasound (Active Comparator): Therapeutic ultrasound applied for a period of 5 minutes to the most painful region of the neck, then a second 5 minute dose at the most painful region of the upper extremity
  Interventions: Device: Therapeutic Ultrasound
- Soft Tissue Mobilization (Experimental): Passive soft tissue mobilization to the neck and upper extremity
  Interventions: Other: Soft Tissue Mobilization

INTERVENTIONS:
Other: Soft Tissue Mobilization — Patients in the STM group received treatment in supine, with their head resting on one pillow and the involved UE positioned in abduction and external rotation to preload the neural structures of the upper limb. Manual pressure was applied to the soft tissues of the upper quadrant in a deep, stroking manner with the intention to improve the mobility of the soft tissues surrounding the pathway of the neural structures of the upper limb as well as any tender or tight tissues. The therapist spent approximately 7 minutes on the neck and scapular region, 4 minutes on the upper arm, and 4 minutes on the forearm and hand. The therapist was allowed to vary the time spent on each region according to his/her assessment of the patient's condition. The procedure lasted a total of 15 minutes.
  Arms: Soft Tissue Mobilization
Device: Therapeutic Ultrasound — Patients received therapeutic US applied for a period of 5 minutes to the most painful region of the neck, then a second 5-minute dose at the most painful region of the upper extremity. The US dose was 0.5 w/cm2, with sonation time 50% and frequency 1 MHz.40,52 The patient lay supine with the hand of the involved upper extremity placed on the abdomen and the elbow supported on a pillow. The two US doses and interaction time with the patient lasted a total of 15 minutes in an attempt to have equal patient/therapist contact between the two groups.
  Arms: Therapeutic Ultrasound

SUMMARY:
The purpose of this study is to investigate effects of soft tissue mobilization versus therapeutic ultrasound in subjects with neck and arm pain who demonstrate neural mechanical sensitivity.

DETAILED DESCRIPTION:
To investigate the immediate effects of soft tissue mobilization (STM) versus therapeutic ultrasound (US) in patients with neck and arm pain who demonstrate neural mechanical sensitivity. Twenty-three patients with neck and arm pain and a positive upper limb neurodynamic test (ULNT) were randomly assigned to receive STM or therapeutic US during a single session. Outcome measures were collected immediately before and after treatment, and at 2-4 day follow-up. Primary outcomes were the Global Rating of Change (GROC), range of motion (ROM) during the ULNT, and pain rating during the ULNT. Secondary measures included the Neck Disability Index (NDI), Patient-Specific Functional Scale (PSFS), Numeric Pain Rating Scale (NPRS), and active range of shoulder abduction motion combined with the wrist neutral or wrist extension.

ELIGIBILITY:
Inclusion Criteria:

1. Active movement dysfunction that could be related to mechanical sensitivity of the neural structures of the upper limb. (i.e. painful shoulder abduction with elbow extension that is limited more when the wrist is extended than when the wrist is in neutral.)
2. Positive response to upper limb neural provocation testing (ULNT 1) (see description below for details)
3. Tenderness to palpation over the cervical nerve trunks, brachial plexus, or along the median nerve.
4. Tender points or taut bands in the muscles of the upper quadrant including the scalenes, cervical paraspinals, trapezius, deltoid, pectoralis major or minor, rotator cuff, biceps, triceps, coracobrachialis, brachialis, radiobrachialis, pronator teres, supinator, forearm extensor, forearm flexor, pronator quadratus, and hand intrinsic muscles.

Exclusion Criteria:

1. Red flags noted in the medical screening questionnaire such as tumor, fracture, history of metabolic disease, prolonged history of corticosteroid use.
2. Signs of central nervous system involvement such as hyper-reflexia (exaggerated response to deep tendon reflex testing), unsteadiness during gait, ataxia, disturbed vision, nystagmus, altered taste, positive Babinski's or Hoffman's reflexes.
3. Cervical spine surgery within the last 3 months.
4. Litigation associated with their neck and/or upper limb pain.
5. Insufficient English language skills to complete the questionnaires and follow-up instructions.
6. Inability to complete the treatment and follow-up schedule.
7. Current pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Costello, PT, DSc, Principal Investigator — Rocky Mountain University Health Sciences; Emilio j Puentedura, PT, DPT, PhD, Study Director — UNLV

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2009 and June 2012 consecutive patients with neck and arm pain presenting to Cayuga Medical Center's Physical Therapy Department were screened for eligibility criteria
Pre-assignment Details: Patients were excluded if they exhibited Red flags in the medical screening questionnaire such as tumor, fracture; had signs of CNS involvement such as hyper-reflexia, ataxia, nystagmus, etc. Cervical spine surgery within 3 months. Litigation, insufficient English language skills, inability to complete study schedule, or were pregnant.
Groups:
- Therapeutic Ultrasound: Therapeutic ultrasound applied for a period of 5 minutes to the most painful region of the neck, then a second 5 minute dose at the most painful region of the upper extremity
  Therapeutic Ultrasound
- Soft Tissue Mobilization: Passive soft tissue mobilization to the neck and upper extremity
  Soft Tissue Mobilization
Period: Overall Study
Arm/Group | Therapeutic Ultrasound | Soft Tissue Mobilization
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapeutic Ultrasound | Soft Tissue Mobilization | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.00 (10.42) | 46.25 (10.42) | 44.22 (10.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Upper Limb Neurodynamic Tesnion (UNLT) Range of Motion
Time Frame: up to 2-4 day follow up
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Therapeutic Ultrasound | Soft Tissue Mobilization
Number analyzed (Participants) | 11 | 12
degrees | 4.60 [-0.60 to 9.80] | 16.00 [9.88 to 22.12]

2. Primary Outcome: Numeric Pain Rating Scale
Description: Measures perceived level of pain on a scale from 0 to 10, where 0 indicates 'no pain' and 10 indicates 'worst imaginable pain'. Therefore, lower scores are better. Outcome results are given and mean changes from pre to post interventions, therefore, a negative value indicates improvement.
Time Frame: up to 2-4 day follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Therapeutic Ultrasound | Soft Tissue Mobilization
Number analyzed (Participants) | 11 | 12
units on a scale | -0.80 [-2.18 to 0.58] | -1.31 [-2.10 to -0.51]

3. Secondary Outcome: Neck Disability Index
Description: Measure of perceived disability on a scale of 0 to 50, where 0 indicates no disability and 50 indicates maximum disability. Therefore, lower scores are better. Outcome results are given and mean changes from pre to post interventions, therefore, a negative value indicates improvement.
Time Frame: 2-4 day follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Therapeutic Ultrasound | Soft Tissue Mobilization
Number analyzed (Participants) | 11 | 12
units on a scale | -1.20 [-5.63 to 3.23] | -6.00 [-12.55 to 0.55]

4. Secondary Outcome: Patient Specific Functional Scale
Description: Perceived ability to perform specific activities on a scale of 0 to 30, where 0 indicates complete inability to perform and 30 indicates able to perform activity at the same level as before injury or problem. Therefore higher scores are better. Outcome results are given and mean changes from pre to post interventions, therefore, a positive value indicates improvement.
Time Frame: at 2-4 day follow up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Therapeutic Ultrasound | Soft Tissue Mobilization
Number analyzed (Participants) | 11 | 12
units on a scale | 0.30 [-0.16 to 0.76] | 1.67 [0.80 to 2.53]

ADVERSE EVENTS:
Time Frame: Baseline to 2 - 4 days follow up
Arm/Group | Therapeutic Ultrasound | Soft Tissue Mobilization
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes